CLINICAL TRIAL: NCT05294770
Title: Efficacy of a Very Low Calorie Diet or a Hypocaloric Mediterranean Diet on Albuminuria and Renal Function in Patients With Obesity-related Glomerulopathy: a Randomized Clinical Trial
Brief Title: Dietary Intervention in Obesity-related Glomerulopathy
Acronym: ORG-VLCD-2022
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORG-VLCD-2022
Record Dates: First submitted 2022-02-01; First posted 2022-03-24 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-01

CONDITIONS: Obesity; Glomerulopathy
Keywords: Albuminuria; Obesity; kidney function; diet; elastography; weight loss
MeSH Terms: conditions — Obesity; Albuminuria; Weight Loss

STUDY DESIGN:
Masking Description: Patients will be randomized in a 1:1 ratio
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Very Low Calorie Diet (VLCD) (Experimental): Patients randomized to this group will receive a VLCD, which consists of a replacement diet based on a liquid enteral formula (46% carbohydrates, 19% fat and 32% protein; 654 Kcal/day): OPTISOURCE® PLUS, taken as 3 shakes a day. In addition, participants may consume 2 pieces of fruit/day (about 250 g/day) and up to 300 g/day of non-starchy vegetables according to the list of foods that will be provided to patients; this will constitute a total daily energy intake of about 800 Kcal. In addition, protein intake (0.8 to 1.3 g/kg/day of adjusted weight) will be adjusted by adding Resource® Instant Protein individually, depending on the anthropometry and the renal function of the patients (to preserve fat free mass, whose loss has been correlated with subsequent weight recovery)
  Interventions: Other: Optisource® Plus: Very Low Calorie Diet treatment
- Hypocaloric Mediterranean diet (Active Comparator): Randomized participants in this group will be recommended to follow a Mediterranean Diet, based on the use of olive oil as the main source of visible fat and regular consumption of vegetables (≥2 servings/day), fruits (≥3 servings/day), legumes (≥3 servings/week) and fish (≥3 times a week), reducing the consumption of red meat or sausages (<2 times a week) and eliminating the consumption of sugary drinks, pastries or industrial pastries. In this Mediterranean Diet, an energy restriction of 30% of the estimated energy needs (Harris-Benedict equation) will be established.
  Interventions: Other: Hypocaloric Mediterranean Diet

INTERVENTIONS:
Other: Optisource® Plus: Very Low Calorie Diet treatment — Patients randomized to this group will receive a VLCD, which consists of a replacement diet based on a liquid enteral formula (46% carbohydrates, 19% fat and 32% protein; 654 Kcal/day): OPTISOURCE® PLUS, taken as 3 shakes a day. In addition, participants may consume 2 pieces of fruit/day (about 250 g/day) and up to 300 g/day of non-starchy vegetables according to the list of foods that will be provided to patients; this will constitute a total daily energy intake of about 800 Kcal. In addition, protein intake (0.8 to 1.3 g/kg/day of adjusted weight) will be adjusted by adding Resource® Instant Protein individually, depending on the anthropometry and the renal function of the patients (to preserve fat free mass, whose loss has been correlated with subsequent weight recovery)
  Arms: Very Low Calorie Diet (VLCD)
Other: Hypocaloric Mediterranean Diet — Randomized participants in this group will be recommended to follow a Mediterranean Diet, based on the use of olive oil as the main source of visible fat and regular consumption of vegetables (≥2 servings/day), fruits (≥3 servings/day), legumes (≥3 servings/week) and fish (≥3 times a week), reducing the consumption of red meat or sausages (<2 times a week) and eliminating the consumption of sugary drinks, pastries or industrial pastries. In this Mediterranean Diet, an energy restriction of 30% of the estimated energy needs (Harris-Benedict equation) will be established.
  Arms: Hypocaloric Mediterranean diet

SUMMARY:
Obesity-related glomerulopathy (ORG) is a silent comorbidity associated with obesity whose incidence is increasing in parallel to the obesity epidemic. ORG is associated with serious health consequences including chronic kidney disease, end-stage renal disease, and increased mortality. Unfortunately, ORG has an absence of targeted therapy (except for the use of drugs blocking the renin-angiotensin system), and therefore the prognosis of this disease may be seriously compromised. Some previous studies have shown that weight loss could be effective to decrease albuminuria and reduce the declining in kidney function in subject with obesity. In line with this, in this study the investigators will evaluate the efficacy of two different dietary strategies for ORG, given the current lack of therapies for this condition. Thus, the investigators will conduct an open-label randomized controlled trial comparing a hypocaloric Mediterranean diet with a very-low calorie diet (VLCD), evaluating the efficacy on albuminuria reduction and changes in renal function. Also, the investigators will assess changes on body composition, blood pressure, markers of renal damage and inflammation, gut microbiota, and on renal ultrasound elastography.

DETAILED DESCRIPTION:
Our hypothesis is that a dietary strategy based on a very low calorie diet (VLCD) will produce a greater reduction in albuminuria than a hypocaloric Mediterranean diet in subjects with ORG. This improvement will be achieved through weight loss and changes in body composition, the reduction of blood pressure, the decrease in inflammatory, tubular and podocyte damage markers, modifications in adipokine concentrations, changes in the intestinal microbiota and in renal elastography.

The main objective of this clinical trial is to evaluate which dietary strategy (VLCD diet or Mediterranean hypocaloric diet) is more effective in reducing albuminuria and preserving renal function in patients with ORG.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 30 kg/m2
* Albuminuria ≥ 150 mg/g
* eGFR ≥ 30 ml/min/1,73 m²
* Informed consent signed
* All patients should receive a stable dose of ACE inhibitors or ARBs for at least 4 weeks prior to randomization. Before randomization; A stable dose will be considered to be the maximum dose indicated in the drug's SmPC or a dose that is not associated with unacceptable side effects in the patient.

Exclusion Criteria:

* Previous diagnosis of diabetes mellitus (defined by HbA1c ≥ 6.5% or baseline blood glucose ≥126 mg / dl or blood glucose 2 hours after oral glucose overload ≥200 mg / dl).
* Treatment with oral hypoglycemic agents, insulin or GLP-1 receptor agonists.
* Active cancer
* History of liver tumor or acute or chronic liver diseases with impaired liver function: total bilirubin levels> 2.0 mg / dL or AST levels three times higher than the upper limit of normal.
* Established cardiovascular disease (stroke, acute myocardial infarction, cardiac revascularization).
* Uncontrolled hypertension (systolic blood pressure> 180 mmHg or diastolic blood pressure> 110 mmHg) despite adequate antihypertensive treatment.
* Infection with HIV, HBV, HCV or other infection that can lead to secondary glomerular disease
* Suspicion of primary glomerulopathy (except GAO).
* Evidence of drug or alcohol abuse.
* Serious underlying conditions that, in the opinion of the investigators, could affect the patient's ability to participate in the study.
* Limited life expectancy (<12 months).
* Pregnancy or breastfeeding.
* Impossibility of following the indicated diet.
* Inability to follow scheduled visits.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-18 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Changes in albuminuria | From baseline to 6 months
  Albuminuria in mg/g

SECONDARY OUTCOMES:
Changes in glomerular filtration (kidney function) | From baseline to 6 months
  Calculated with the formula CKD-EPI and measured in ml/min/1,73 m2
Cystatin C levels (kidney function) | From baseline to 6 months
  Cystatin C in ng/ml
BMI (body mass index) | From baseline to 6 months
  kg/m2
Changes in total body water (TBW) | From baseline to 6 months
  Measured in liters
Changes in extracellular water (ECW) | From baseline to 6 months
  Measured in liters
Changes in intracellular water (ICW) | From baseline to 6 months
  Measured in liters
Changes in fat free mass (FFM) | From baseline to 6 months
  Measured in kilograms
Changes in fat free mass index (FFMI) | From baseline to 6 months
  Measured in Kg/m2
Changes in fat mass (FM) | From baseline to 6 months
  Measured in Kilograms
Changes in fat mass index (FMI) | From baseline to 6 months
  Measured in Kg/m2
Changes in body cell mass (BCM) | From baseline to 6 months
  Measured in kilograms
Changes in body cell mass index (BCMI) | From baseline to 6 months
  Measured in Kg/m2
Changes in appendicular skeletal muscle mass (ASMM) | From baseline to 6 months
  Measured in kilograms
Changes in blood pressure | From baseline to 6 months
  We will perform a 24-hour Ambulatory Blood Pressure Measurement (ABPM) with the SpaceLab © OnTrak meter (Spacelabs Healthcare, Washington, USA), the newest ABPM meter from this recognized manufacturer. This ABPM meter is a clinically validated device with high precision and reliability.
Changes in inflammatory biomarkers (assess kidney failure) | From baseline to 6 months
  Measured as Fetuin A, FGF-21 and TGF-β1 by ELISA (ng/ml)
Changes in tubular and podocyte damage markers (assess kidney failure) | From baseline to 6 months
  Measured as KIM-1 y NGAL by ELISA (ng/ml)
Changes in adipokines | From baseline to 6 months
  Measured as leptin, adiponectin and resistin by ELISA (ng/ml)
Modifications in gut microbiota richness and diversity | From baseline to 6 months
  Differences in α- and β-diversities between study groups will be analyzed with the open-source Quantitative Insights into Microbial Ecology (QIIME2) software, through the diversity plugin
Modifications in gut microbiota abundance and composition | From baseline to 6 months
  Differences between the study groups at different taxa levels (phyla, family, genus and species) will be evaluated with the QIIME2 software
Modifications in gut microbiota functionality | From baseline to 6 months
  We will evaluate the differences between sudy groups in microbial functions, analyzed with the Phylogenetic Investigation of Communities by Reconstruction of Unobserved States (PICRUSt2) software, within the QIIME2 environment
Modifications in shear-wave renal elastography | From baseline to 6 months
  Changes in kilopascals (kPA) in renal sinus

CONTACTS AND LOCATIONS:
Overall Officials: José Carlos Fernández García, MD, PhD., Principal Investigator — Hospital Regional Universitario de Málaga - FIMABIS
Locations (1):
- Hospital Regional Universitario de Málaga., Málaga, Spain